CLINICAL TRIAL: NCT06822608
Title: Evaluation of a Fixed Combination of Dexpanthenol and Hyaluronic Acid Preservative-free Eye Drops on Corneal Epithelialization After Trans Epithelial PRK: a Prospective, Contralateral, Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Evaluation of Dexpanthenol and Hyaluronic Acid Eye Drops on Corneal Epithelialization After Trans Epithelial PRK
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Katsimpras Marios, Principal Investigator, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT72975
Record Dates: First submitted 2024-09-27; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Corneal Epithelial Wound Healing
Keywords: epithelial defect; re-epithelialization; reepithelialization; dexpanthenol; trans - PRK; contrallateral study; double-blinded study; prospective study; corneal healing; corneal epithelium healing
MeSH Terms: interventions — dexpanthenol

STUDY DESIGN:
Intervention Model Description: This is a contralateral, randomized, double-blind, placebo-controlled (HA) trial.
  One eye of each patient, randomly determined, will be assigned to receive artificial tears containing a combination of dexpanthenol-hyaluronic acid (study group) while the fellow eye will receive Placebo / identical combination containing the same ingredients and hyaluronic acid without dexpanthenol (control group). The drops will be applied hourly postoperatively, starting one hour after the surgery. The subject will participate in 1 preoperative visit, 1 postoperatively visit and following daily visits until complete reepithelialization of both eyes or day 7 postoperatively. Researchers will compare the epithelialization between the two eyes.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fixed combination of dexpanthenol and hyaluronic acid eye drops (Active Comparator): Subjects will receive 1 drop of a fixed combination of dexpanthenol and hyaluronic acid preservative-free eye artificial tears eye drops (DexHA) hourly during the day, but at least 12 times a day, until complete reepithelialization
  Interventions: Drug: dexpanthenol and hyaluronic acid preservative-free eye artificial tears eye drops
- Placebo eye drops (Placebo Comparator): Subjects will receive 1 drop of a hyaluronic acid preservative-free eye artificial tears eye drops (HA) as PLACEBO hourly during the day, but at least 12 times a day, until complete reepithelialization
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: dexpanthenol and hyaluronic acid preservative-free eye artificial tears eye drops — Subjects will receive 1 drop of a hyaluronic acid preservative-free eye artificial tears eye drops (HA) as PLACEBO hourly during the day, but at least 12 times a day, until complete reepithelialization. Composition: 1 ml contains Sodium Hyaluronate 0.15 %, Sodium Chloride, Sodium Citrate, Citric Acid, Water for Injections Dosage Form: Single-dose container (0.5 mL)
  Arms: Fixed combination of dexpanthenol and hyaluronic acid eye drops
Drug: Placebo — Subjects will receive 1 drop of a hyaluronic acid preservative-free eye artificial tears eye drops (HA) as PLACEBO hourly during the day, but at least 12 times a day, until complete reepithelialization. Composition: 1 ml contains Sodium Hyaluronate 0.15 %, Sodium Chloride, Sodium Citrate, Citric Acid, Water for Injections Dosage Form: Single-dose container (0.5 mL)
  Arms: Placebo eye drops

SUMMARY:
The aim of this prospective, contralateral, randomized, double-blind, placebo-controlled study is the evaluation of the performance of a fixed combination of dexpanthenol and hyaluronic acid preservative-free eye artificial tears eye drops, in corneal wound healing after trans epithelial photorefractive keratectomy. One eye of each patient, randomly determined, will be assigned to receive artificial tears containing a combination of dexpanthenol-hyaluronic acid (study group) while the fellow eye will receive Placebo / identical combination containing the same ingredients and hyaluronic acid without dexpanthenol (control group). The drops will be applied hourly postoperatively, starting one hour after the surgery. All subjects will be treated until the day of complete reepithelialization or a maximum of 7 days postoperatively. Researchers will compare the epithelialization between the two eyes. The primary endpoint is the time to reepithelialization.The secondary endpoints are the intra-individual differences measured in each eye in terms of epithelial defect size in each visit, subjective evaluation of pain (discomfort) and subjective evaluation of vision.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged ≥ 18
* Bilateral trans PRK for the correction of myopia using the Schwind Amaris 1050RS laser at the same treatment zone (6.5mm)
* Signed written informed consent Ability and willingness to participate in all examinations

Exclusion Criteria:

* Known hypersensitivity or intolerance to any component of the product
* Previous refractive surgery
* Myopic refractive error higher than 8.00 diopters (D)
* Anisometropia higher than 2.00 D
* Ocular or systemic disease that could affect epithelial healing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Time to reepithelialization. | From the day of the surgery until complete reepithelialization of both eyes or day 7 postoperatively.
  The primary endpoint is the time to reepithelialization. Slitlamp biomicroscopy will be preformed to evaluate the integrity of the corneal media and objectively assess epithelial healing with the use of fluoroscein staining. Α record of the time needed until no staining is present will be made.

SECONDARY OUTCOMES:
Epithelial defect size in each visit | From the day of the surgery until complete reepithelialization of both eyes or day 7 postoperatively.
  Epithelial defect size at each visit measured by slitlamp biomicroscopy The integrity of the corneal media is calculated from the remaining area (A) of the epithelial defects using the following equation: A=π {(α +b) /4}2 where a is the shortest dimension of the defect and b is the longest dimension.
Subjective evaluation of pain (discomfort) | From the day of the surgery until complete reepithelialization of both eyes or day 7 postoperatively.
  Pain scores will be evaluated using a questionnaire on a scale of 0 to 4 as follows:
  * 0 as no discomfort or pain
  * 1 as mild discomfort
  * 2 as moderate burning pain
  * 3 as burning pain requiring oral medication (nimesulide 100 mg)
  * 4 as severe constant or sharp pain not mitigated with oral medication.
Subjective evaluation of vision | From the day of the surgery until complete reepithelialization of both eyes or day 7 postoperatively.
  Uncorrected distance visual acuity measured using logMAR ETDRS charts at 4 m

CONTACTS AND LOCATIONS:
Locations (1):
- National and Kapodistrian University of Athens, Athens, Greece, Greece